CLINICAL TRIAL: NCT05860621
Title: Promoting Physical Activity Through Supervised vs Motivational Behavior Change Interventions in Breast Cancer Survivors on Aromatase Inhibitors (PAC-WOMAN): A 3-arm Pragmatic Randomized Controlled Trial
Brief Title: Promoting Physical Activity in Breast Cancer Survivors on Aromatase Inhibitors
Acronym: PAC-WOMAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo Lusófona (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); Faculdade de Motricidade Humana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PAC-WOMAN; PTDC/SAU-DES/2865/2020 (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia)
Record Dates: First submitted 2023-04-20; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer Female; Hormone-receptor-positive Breast Cancer

STUDY DESIGN:
Intervention Model Description: A 3-arm randomized controlled trial, involving a 4-month intervention period and a 12-month follow-up, will be implemented to compare: 1) a brief PA counseling intervention; 2) a structured exercise program; and 3) a waiting-list control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brief Physical Activity Counselling (Experimental): The brief physical activity counselling (PAC) group will receive a group-based, light-touch, motivational counselling program to promote physical activity.
  Interventions: Behavioral: Brief Physical Activity Counselling
- Structured Exercise Program (Experimental): The structured exercise group will receive a group-based supervised multi-component exercise program, with progressive intensity.
  Interventions: Behavioral: Structured Exercise Program
- Waitlist control (No Intervention): Patients allocated to the control group (i.e., waiting list) will keep daily routines and standard medical care. At the end of the study, the control group will be offered the structured exercise program.

INTERVENTIONS:
Behavioral: Brief Physical Activity Counselling — The brief physical activity counselling program will comprise 8 sessions (120 minutes each), every fifteen days, addressing the following themes: reasons to change, an introduction to the PAC-WOMAN program and principles, types of physical activity and their benefits, strategies on how to become more active and less sedentary, how to safely practice exercise at home, the importance of social support for doing more physical activity, barriers and facilitators for becoming more active, development of coping plans and strategies to overcome those barriers, establishing SMART goals, self-monitoring, medical aspects related to symptom management in breast cancer survivors, body image and self-acceptance, sharing experiences with role models, and re-evaluating action plans. It will be delivered in a need-supportive interpersonal climate, according to Self-Determination Theory principles.
  Arms: Brief Physical Activity Counselling
Behavioral: Structured Exercise Program — The structured exercise program was informed by the most recent guidelines for exercise prescription and safe practice in cancer populations. A supervised program of 32 sessions (over 4 months), lasting 90 min each, and taking place twice a week, was developed. The program combines aerobic, strength and mobility exercises, and is organized in four mesocycles, with progressive intensity, always adapted according to participants' initial assessments and evolution throughout the weeks. Once every 15 days, a thematic group class will be offered to participants, so that they can experiment and discover new physical activities, and more easily maintain regular practice in the future.
  Arms: Structured Exercise Program

SUMMARY:
Aromatase inhibitors (AI) are frequently used to treat hormone-receptor-positive breast cancer, but they have multiple adverse effects (eg, arthralgia), resulting in premature therapy discontinuation/switch. Physical activity (PA) can attenuate these negative effects and improve quality of life (QoL). However, most cancer survivors fail to perform/sustain adequate PA levels, especially in the long-term. Theory-based interventions, using evidence-based behavior change techniques, aimed at promoting long-term behavior change in breast cancer survivors are effective, but remain scarce and fail to promote self-regulatory skills and better-quality motivations associated with sustained PA adoption.

PAC-WOMAN will test the long-term effectiveness and cost-effectiveness of two state of the art, group-based interventions encouraging sustained changes in PA, sedentary behavior, and QoL. Additional aims include examining the impact of both interventions on secondary outcomes (eg, body composition, physical function), and key moderators/mediators of short and long-term changes in primary outcomes. A 3-arm pragmatic randomized controlled trial, involving a 4-month intervention and a 12-month follow-up, will be implemented, in a real exercise setting, to compare: 1) brief PA counseling/motivational intervention; 2) structured exercise program vs. waiting-list control group. Study recruitment goal is 122 hormone-receptor-positive breast cancer survivors (stage I-III), on AI therapy (post-primary treatment completion) ≥1 month, performance status 0-1. Outcome measures will be obtained at baseline, 4 months (i.e., post-intervention), 10 and 16 months. Process evaluation, analyzing implementation determinants, will also be conducted.

PAC-WOMAN is expected to have a relevant impact on participants PA and QoL, and on the improvement of interventions designed to promote sustained adherence to active lifestyle behaviors, facilitating its translation to community settings.

DETAILED DESCRIPTION:
Aromatase inhibitors (AI) are frequently used to treat hormone-receptor-positive breast cancer, but they have multiple adverse effects (eg, osteoporosis, arthralgia), resulting in premature therapy discontinuation/switch. Physical activity (PA) is safe and should be an integral and continuous part of care for all individuals diagnosed with cancer. There is compelling evidence suggesting that PA plays an important role in improving longevity among cancer survivors. PA effectively ameliorates short- and long-term adverse effects of cancer therapies (eg, comorbid conditions, improves physical fitness and function, attenuates cancer-related fatigue, enhances body image and quality of life (QoL), and decreases cancer recurrence and mortality. PA also allows women to benefit from endocrine therapy while being protected against the related risk of osteoporosis, fracture, and ultimately cancer recurrence or death. Thus, PA in breast cancer survivors, and specifically among women on AIs, is paramount to improve health outcomes, QoL, and prevent therapy discontinuation. However, most cancer survivors fail to meet established guidelines for PA.

Theory-based interventions, using evidence-based behavior change techniques, aimed at promoting long-term health behavior change in breast cancer survivors are effective, but remain scarce and predominantly focused on short-term adherence/outcomes. Also, most interventions fail to provide validated self-regulatory tools or explore meaningful links between PA and patients' values and life aspirations to foster lasting behavior changes. Prior research has shown that internal (better quality) forms of motivation play an important role in PA and behavior sustainability, suggesting that self-determination theory (SDT) can be a valid framework to promote sustained adherence to PA. A need-supportive intervention climate enhances people's wellbeing and their ability to self-regulate and sustain behavior changes. Finally, skills such as self-monitoring, goal setting or action planning have also been identified as important mediators of long-term PA and as core features of effective behavior change/maintenance interventions in breast cancer survivors.

In sum, although regular PA is a promising and safe way of helping cancer survivors navigate their disease, alleviating the growing pressure on the health care system, most cancer survivors do not meet the recommended PA doses. It is a goal of this project to overcome the abovementioned shortcomings, by testing an intervention model informed by solid evidence and a robust theoretical rationale (SDT), provided by qualified exercise professionals, which appear to add value to the treatment process, improving the therapeutic effect and safety of the exercise practice.

PAC-WOMAN will test the long-term effectiveness and cost-effectiveness of two 4-month group-based interventions aimed at promoting sustained changes in PA, sedentary behavior, and QoL. Additional aims include examining the impact of both interventions on secondary outcomes (eg, body composition, physical function), and key moderators and mediators of short and long-term changes in primary outcomes. A 3-arm randomized controlled trial, involving a 4-month intervention period and a 12-month follow-up, will be implemented to compare: 1) a brief PA counseling intervention; 2) a structured exercise program; and 3) a. waiting-list control group. Study recruitment goal is 122 breast cancer survivors with hormone-receptor-positive breast cancer (stage I-III), on AI therapy (post-primary treatment completion) for at least 1 month, ECOG performance status 0-1. Outcome measures will be obtained at baseline, 4 months (i.e., post-intervention), 10 and 16 months. Process evaluation, analyzing implementation determinants, will also be conducted.

PAC-WOMAN is expected to have a relevant impact on the improvement of interventions designed to promote sustained adherence to active lifestyle behaviors and facilitate its translation to community settings.

ELIGIBILITY:
Inclusion Criteria:

1. post-menopausal women, below 70 years old;
2. histologically confirmed hormone-receptor-positive breast cancer (stage I, II, III);
3. having initiated aromatase inhibitor hormonal therapy following the primary treatment (surgery, radiotherapy, chemotherapy, etc.), at least 1 month before being enrolled;
4. ECOG-Performance Status 0-1.

Exclusion Criteria:

1. evidence of stage IV cancer or synchronous tumors;
2. uncontrolled hypertension, cardiac or pulmonary disease;
3. contraindications to exercise training according to the assistant doctor;
4. inability to provide informed consent;
5. expected inability to fulfill the proposed schedule.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Physical activity on Actigraph GT9X accelerometers at 16 months | baseline and 16 months
  Accelerometers Actigraph GT9X will be worn in the wrist for 7 days to assess the amount of activity expressed as minutes per day spent in different intensities (sedentary, light, moderate, vigorous).
Change from baseline in Physical activity on Actigraph GT9X accelerometers at 4 months | baseline and 4 months
  Accelerometers Actigraph GT9X will be worn in the wrist for 7 days to assess the amount of activity expressed as minutes per day spent in different intensities (sedentary, light, moderate, vigorous).
Change from baseline in Physical activity on Actigraph GT9X accelerometers at 10 months | baseline and 10 months
  Accelerometers Actigraph GT9X will be worn in the wrist for 7 days to assess the amount of activity expressed as minutes per day spent in different intensities (sedentary, light, moderate, vigorous).
Change from baseline in self-reported physical activity on International Physical Activity Questionnaire (IPAQ-sf) at 16 months | baseline and 16 months
  The 9-item IPAQ-sf measures the weekly frequency and duration of PA across three specific intensities (i.e., light, moderate, and vigorous), and time spent sitting during week and weekend days. Scores for weekly minutes of total physical activity, and discriminated by intensity, will be obtained. Total minutes of sitting time will be also obtained.
Change from baseline in self-reported physical activity on International Physical Activity Questionnaire (IPAQ-sf) at 4 months | baseline and 4 months
  The 9-item IPAQ-sf measures the weekly frequency and duration of PA across three specific intensities (i.e., light, moderate, and vigorous), and time spent sitting during week and weekend days. Scores for weekly minutes of total physical activity, and discriminated by intensity, will be obtained. Total minutes of sitting time will be also obtained.
Change from baseline in self-reported physical activity on International Physical Activity Questionnaire (IPAQ-sf) at 10 months | baseline and 10 months
  The 9-item IPAQ-sf measures the weekly frequency and duration of PA across three specific intensities (i.e., light, moderate, and vigorous), and time spent sitting during week and weekend days. Scores for weekly minutes of total physical activity, and discriminated by intensity, will be obtained. Total minutes of sitting time will be also obtained.
Change from baseline in cancer-related quality of fife on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) and its breast cancer module (EORTC-BR23) at 16 months | baseline and 16 months
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) and its breast cancer module (EORTC QLQ-BR23). Five items specifically related to joint, bone, and muscle pain/discomfort, derived from the new EORTC QLQ-BR45, were added provided the specificity of aromatase inhibitors' side effects. Scores generally range from 1 to 4. Higher scores generally reflect worse quality of life.
Change from baseline in cancer-related quality of fife on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) and its breast cancer module (EORTC-BR23) at 4 months | baseline and 4 months
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) and its breast cancer module (EORTC QLQ-BR23). Five items specifically related to joint, bone, and muscle pain/discomfort, derived from the new EORTC QLQ-BR45, were added provided the specificity of aromatase inhibitors' side effects. Scores generally range from 1 to 4. Higher scores generally reflect worse quality of life.
Change from baseline in cancer-related quality of fife on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) and its breast cancer module (EORTC-BR23) at 10 months | baseline and 10 months
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) and its breast cancer module (EORTC QLQ-BR23). Five items specifically related to joint, bone, and muscle pain/discomfort, derived from the new EORTC QLQ-BR45, were added provided the specificity of aromatase inhibitors' side effects. Scores generally range from 1 to 4. Higher scores generally reflect worse quality of life.
Healthcare Use | 6-month after the end of the intervention
  Healthcare use will be assessed by phone interview 6 months after ending the intervention period. Data will be collected on healthcare resources use during the study period, namely number and type of consultations, drugs, medical tests and exams, in-patient stays and day care sessions. Absenteeism will be assessed using participants' reports of their number of absence days or percentage of normal working hours worked, valued at patients' hourly wage. These resources will then be valued using usual official sources.

SECONDARY OUTCOMES:
Change from baseline in body composition on bioelectrical impedance at 16 months | baseline, 4 months (intervention's end), 10 and 16 months
  Body composition will be assessed using Bioelectrical Impedance, under standardized conditions, by experienced technicians and oversaw by the research team.
Change from baseline in body composition on bioelectrical impedance at 4 months | baseline and 4 months
  Body composition will be assessed using Bioelectrical Impedance, under standardized conditions, by experienced technicians and oversaw by the research team.
Change from baseline in body composition on bioelectrical impedance at 10 months | baseline and 10 months
  Body composition will be assessed using Bioelectrical Impedance, under standardized conditions, by experienced technicians and oversaw by the research team.
Change from baseline in body mass index (BMI) at 16 months | baseline and 16 months
  Body mass index (BMI in kilograms per square meter) will be calculated from weight (kg; measured with a digital SECA scale) and height (m; measured with a balance-mounted stadiometer). BMI = weight/(height*height).
Change from baseline in body mass index (BMI) at 4 months | baseline and 4 months
  Body mass index (BMI in kilograms per square meter) will be calculated from weight (kg; measured with a digital SECA scale) and height (m; measured with a balance-mounted stadiometer). BMI = weight/(height*height).
Change from baseline in body mass index (BMI) at 10 months | baseline and 10 months
  Body mass index (BMI in kilograms per square meter) will be calculated from weight (kg; measured with a digital SECA scale) and height (m; measured with a balance-mounted stadiometer). BMI = weight/(height*height).
Change from baseline in cardio-respiratory fitness at 16 months | baseline and 16 months
  Cardiorespiratory fitness will be assessed with a submaximal, 8-min, single-stage walking test on a treadmill, involving a 4-min warming up at a self-selected speed, at 50-70% of the individual's age-predicted maximum heart rate, and 4 additional minutes at a 5%-increased workload. The steady-state heart rate at this workload and the treadmill speed, together with participants' age and gender, will be used to estimate VO2max.
Change from baseline in cardio-respiratory fitness at 4 months | baseline and 4 months
  Cardiorespiratory fitness will be assessed with a submaximal, 8-min, single-stage walking test on a treadmill, involving a 4-min warming up at a self-selected speed, at 50-70% of the individual's age-predicted maximum heart rate, and 4 additional minutes at a 5%-increased workload. The steady-state heart rate at this workload and the treadmill speed, together with participants' age and gender, will be used to estimate VO2max.
Change from baseline in cardio-respiratory fitness at 10 months | baseline and 10 months
  Cardiorespiratory fitness will be assessed with a submaximal, 8-min, single-stage walking test on a treadmill, involving a 4-min warming up at a self-selected speed, at 50-70% of the individual's age-predicted maximum heart rate, and 4 additional minutes at a 5%-increased workload. The steady-state heart rate at this workload and the treadmill speed, together with participants' age and gender, will be used to estimate VO2max.
Change from baseline in strength at 16 months | baseline and 16 months
  Handgrip strength will be measured with a handgrip dynamometer. Participants will be instructed to hold the handgrip with their maximal strength. Dynamic muscle strength will be determined for chest press, seated row and leg press, using a 10-repetition maximum (10 RM) test. After a standardized warm-up, gradual load increases will be made until the maximum weight lifted through a full range of motion will be recorded as 10 RM.
Change from baseline in strength at 4 months | baseline and 4 months
  Handgrip strength will be measured with a handgrip dynamometer. Participants will be instructed to hold the handgrip with their maximal strength. Dynamic muscle strength will be determined for chest press, seated row and leg press, using a 10-repetition maximum (10 RM) test. After a standardized warm-up, gradual load increases will be made until the maximum weight lifted through a full range of motion will be recorded as 10 RM.
Change from baseline in strength at 10 months | baseline and 10 months
  Handgrip strength will be measured with a handgrip dynamometer. Participants will be instructed to hold the handgrip with their maximal strength. Dynamic muscle strength will be determined for chest press, seated row and leg press, using a 10-repetition maximum (10 RM) test. After a standardized warm-up, gradual load increases will be made until the maximum weight lifted through a full range of motion will be recorded as 10 RM.
Change from baseline in physical function on the Stand on one foot Test at 16 months | baseline and 16 months
  In the Stand on one foot test, participants are instructed to stand on one foot with their eyes open (both sides are tested) for a maximum of 20 seconds and have their time recorded.
Change from baseline in physical function on the Stand on one foot Test at 4 months | baseline and 4 months
  In the Stand on one foot test, participants are instructed to stand on one foot with their eyes open (both sides are tested) for a maximum of 20 seconds and have their time recorded.
Change from baseline in physical function on the Stand on one foot Test at 10 months | baseline and 10 months
  In the Stand on one foot test, participants are instructed to stand on one foot with their eyes open (both sides are tested) for a maximum of 20 seconds and have their time recorded.
Change from baseline in physical function on the Sit to Stand Test at 16 months | baseline and 16 months
  The Sit to Stand Test consists of standing and seating in a chair as many times as possible with arms crossed over the chest in 30 seconds.
Change from baseline in physical function on the Sit to Stand Test at 4 months | baseline and 4 months
  The Sit to Stand Test consists of standing and seating in a chair as many times as possible with arms crossed over the chest in 30 seconds.
Change from baseline in physical function on the Sit to Stand Test at 10 months | baseline and 10 months
  The Sit to Stand Test consists of standing and seating in a chair as many times as possible with arms crossed over the chest in 30 seconds.
Change from baseline in physical function on the Timed up and go Test at 16 months | baseline and 16 months
  The Time Up and Go Test is used to assess mobility by measuring the time a person takes to rise from a chair, walk 2.44 meters, turn around, walk back to the chair, and sit down.
Change from baseline in physical function on the Timed up and go Test at 4 months | baseline and 4 months
  The Time Up and Go Test is used to assess mobility by measuring the time a person takes to rise from a chair, walk 2.44 meters, turn around, walk back to the chair, and sit down.
Change from baseline in physical function on the Timed up and go Test at 10 months | baseline and 10 months
  The Time Up and Go Test is used to assess mobility by measuring the time a person takes to rise from a chair, walk 2.44 meters, turn around, walk back to the chair, and sit down.
Change from baseline in flexibility using angular measures at 16 months | baseline and 16 months
  Angular measures of shoulder flexion and abduction will be measured on both sides using a goniometer.
Change from baseline in flexibility using angular measures at 4 months | baseline and 4 months
  Angular measures of shoulder flexion and abduction will be measured on both sides using a goniometer.
Change from baseline in flexibility using angular measures at 10 months | baseline and 10 months
  Angular measures of shoulder flexion and abduction will be measured on both sides using a goniometer.
Change from baseline in flexibility using linear measures at 16 months | baseline and 16 months
  Linear measures will be measured using the Back Scratch protocol on both shoulders with a SECA measuring tape.
Change from baseline in flexibility using linear measures at 4 months | baseline and 4 months
  Linear measures will be measured using the Back Scratch protocol on both shoulders with a SECA measuring tape.
Change from baseline in flexibility using linear measures at 10 months | baseline and 10 months
  Linear measures will be measured using the Back Scratch protocol on both shoulders with a SECA measuring tape.
Change from baseline in pain severity on the Brief Pain Inventory at 16 months | baseline and 16 months
  Single items of the Brief Pain Inventory (BPI) will be used to assess pain severity "on average" and "right now". Scores range from 0 (no pain) to 10 (the worst pain ever). Higher scores reflect higher pain severity.
Change from baseline in pain severity on the Brief Pain Inventory at 4 months | baseline and 4 months
  Single items of the Brief Pain Inventory (BPI) will be used to assess pain severity "on average" and "right now". Scores range from 0 (no pain) to 10 (the worst pain ever). Higher scores reflect higher pain severity.
Change from baseline in pain severity on the Brief Pain Inventory at 10 months | baseline and 10 months
  Single items of the Brief Pain Inventory (BPI) will be used to assess pain severity "on average" and "right now". Scores range from 0 (no pain) to 10 (the worst pain ever). Higher scores reflect higher pain severity.
Change from baseline in pain interference on the Pain Disability Index at 16 months | baseline and 16 months
  The 7-item Pain Disability Index (PDI) will be used to evaluate the impact and interference of pain on participants' daily activities and functioning (i.e., family and home responsibilities, recreation, social activity, occupation, sexual behavior, self-care, and life-support activities). Scores range from 0 (no incapacity) to 10 (total incapacity). Higher scores reflect higher pain interference with daily activities.
Change from baseline in pain interference on the Pain Disability Index at 4 months | baseline and 4 months
  The 7-item Pain Disability Index (PDI) will be used to evaluate the impact and interference of pain on participants' daily activities and functioning (i.e., family and home responsibilities, recreation, social activity, occupation, sexual behavior, self-care, and life-support activities). Scores range from 0 (no incapacity) to 10 (total incapacity). Higher scores reflect higher pain interference with daily activities.
Change from baseline in pain interference on the Pain Disability Index at 10 months | baseline and 10 months
  The 7-item Pain Disability Index (PDI) will be used to evaluate the impact and interference of pain on participants' daily activities and functioning (i.e., family and home responsibilities, recreation, social activity, occupation, sexual behavior, self-care, and life-support activities). Scores range from 0 (no incapacity) to 10 (total incapacity). Higher scores reflect higher pain interference with daily activities.
Change from baseline in sleep quality on the Pittsburgh Sleep Quality Index at 16 months | baseline and 16 months
  The 19-item Pittsburgh Sleep Quality Index (PSQI) will be used to measure sleep duration (total hours of sleep) and sleep disturbance components of sleep quality (scores range from 0 (no problems to sleep) to 3 (problems > 3 days/week). Higher scores represent poorer sleep quality (less problems) in general. Overall sleep quality is scores from 1 (very bad) to 4 (very good). Higher scores reflect greater sleep quality.
Change from baseline in sleep quality on the Pittsburgh Sleep Quality Index at 4 months | baseline and 4 months
  The 19-item Pittsburgh Sleep Quality Index (PSQI) will be used to measure sleep duration (total hours of sleep) and sleep disturbance components of sleep quality (scores range from 0 (no problems to sleep) to 3 (problems > 3 days/week). Higher scores represent poorer sleep quality (less problems) in general. Overall sleep quality is scores from 1 (very bad) to 4 (very good). Higher scores reflect greater sleep quality.
Change from baseline in sleep quality on the Pittsburgh Sleep Quality Index at 10 months | baseline and 10 months
  The 19-item Pittsburgh Sleep Quality Index (PSQI) will be used to measure sleep duration (total hours of sleep) and sleep disturbance components of sleep quality (scores range from 0 (no problems to sleep) to 3 (problems > 3 days/week). Higher scores represent poorer sleep quality (less problems) in general. Overall sleep quality is scores from 1 (very bad) to 4 (very good). Higher scores reflect greater sleep quality.
Change from baseline in Body Image on the Body Image Scale at 16 months | baseline and 16 months
  The 10-item Body Image Scale (BIS) will be used to assess participants' affective (e.g., feeling self-conscious), behavioral (e.g., difficulty at looking at the naked body), and cognitive (e.g., satisfaction with appearance) dimensions of body image. Scores range from 1 (nothing at all) to 4 (very much). Higher scores reflect poorer body image.
Change from baseline in Body Image on the Body Image Scale at 4 months | baseline and 4 months
  The 10-item Body Image Scale (BIS) will be used to assess participants' affective (e.g., feeling self-conscious), behavioral (e.g., difficulty at looking at the naked body), and cognitive (e.g., satisfaction with appearance) dimensions of body image. Scores range from 1 (nothing at all) to 4 (very much). Higher scores reflect poorer body image.
Change from baseline in Body Image on the Body Image Scale at 10 months | baseline and 10 months
  The 10-item Body Image Scale (BIS) will be used to assess participants' affective (e.g., feeling self-conscious), behavioral (e.g., difficulty at looking at the naked body), and cognitive (e.g., satisfaction with appearance) dimensions of body image. Scores range from 1 (nothing at all) to 4 (very much). Higher scores reflect poorer body image.
Change from baseline in depressive symptoms on the Hospital Anxiety and Depression Scale at 16 months | baseline and 16 months
  The 7-item depression subscale from the Hospital Anxiety and Depression Scale (HADS) will be used to measure depression. Scores range from 1 (no time at all) to 4 (most of the time). Higher scores reflect greater depressive symptoms.
Change from baseline in depressive symptoms on the Hospital Anxiety and Depression Scale at 4 months | baseline and 4 months
  The 7-item depression subscale from the Hospital Anxiety and Depression Scale (HADS) will be used to measure depression. Scores range from 1 (no time at all) to 4 (most of the time). Higher scores reflect greater depressive symptoms.
Change from baseline in depressive symptoms on the Hospital Anxiety and Depression Scale at 10 months | baseline and 10 months
  The 7-item depression subscale from the Hospital Anxiety and Depression Scale (HADS) will be used to measure depression. Scores range from 1 (no time at all) to 4 (most of the time). Higher scores reflect greater depressive symptoms.
Change from baseline in psychological well-being at 16 months | baseline and 16 months
  The various dimensions of psychological well-being will be assessed using 4 items, asking participants to rate their overall satisfaction with life, optimism, and purpose of life and daily activities. Scores range from 1 (not at all) to 10 (completely). Higher scores mean greater psychological well-being and life satisfaction.
Change from baseline in psychological well-being at 4 months | baseline and 4 months
  The various dimensions of psychological well-being will be assessed using 4 items, asking participants to rate their overall satisfaction with life, optimism, and purpose of life and daily activities. Scores range from 1 (not at all) to 10 (completely). Higher scores mean greater psychological well-being and life satisfaction.
Change from baseline in psychological well-being at 10 months | baseline and 10 months
  The various dimensions of psychological well-being will be assessed using 4 items, asking participants to rate their overall satisfaction with life, optimism, and purpose of life and daily activities. Scores range from 1 (not at all) to 10 (completely). Higher scores mean greater psychological well-being and life satisfaction.
Change from baseline in exercise motivations on the Behavioral Regulation in Exercise Questionnaire-3 at 16 months | baseline and 16 months
  The 24-item Behavioral Regulation in Exercise Questionnaire-3 (BREQ-3) will be used to measure the six forms of motivation proposed by self-determination theory - amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic motivation. Scores range from 1 ("Strongly Disagree) to 4 ("Strongly Agree"). Higher scores reflect greater levels of the respective form of motivation.
Change from baseline in exercise motivations on the Behavioral Regulation in Exercise Questionnaire-3 at 4 months | baseline and 4 months
  The 24-item Behavioral Regulation in Exercise Questionnaire-3 (BREQ-3) will be used to measure the six forms of motivation proposed by self-determination theory - amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic motivation. Scores range from 1 ("Strongly Disagree) to 4 ("Strongly Agree"). Higher scores reflect greater levels of the respective form of motivation.
Change from baseline in exercise motivations on the Behavioral Regulation in Exercise Questionnaire-3 at 10 months | baseline and 10 months
  The 24-item Behavioral Regulation in Exercise Questionnaire-3 (BREQ-3) will be used to measure the six forms of motivation proposed by self-determination theory - amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic motivation. Scores range from 1 ("Strongly Disagree) to 4 ("Strongly Agree"). Higher scores reflect greater levels of the respective form of motivation.
Change from baseline in Exercise Needs Satisfaction and Frustration at 16 months | baseline and 16 months
  The 24-item Basic Psychological Need Satisfaction and Frustration Scale (BPNSFS) will be used to assess satisfaction/frustration of the three basic psychological needs (autonomy, competence, and relatedness) for exercise. Scores range from one ("Totally disagree") to five ("Totally agree"). Higher scores mean higher levels of satisfaction/frustration in the respective subscales.
Change from baseline in Exercise Needs Satisfaction and Frustration at 4 months | baseline and 4 months
  The 24-item Basic Psychological Need Satisfaction and Frustration Scale (BPNSFS) will be used to assess satisfaction/frustration of the three basic psychological needs (autonomy, competence, and relatedness) for exercise. Scores range from one ("Totally disagree") to five ("Totally agree"). Higher scores mean higher levels of satisfaction/frustration in the respective subscales.
Change from baseline in Exercise Needs Satisfaction and Frustration at 10 months | baseline and 10 months
  The 24-item Basic Psychological Need Satisfaction and Frustration Scale (BPNSFS) will be used to assess satisfaction/frustration of the three basic psychological needs (autonomy, competence, and relatedness) for exercise. Scores range from one ("Totally disagree") to five ("Totally agree"). Higher scores mean higher levels of satisfaction/frustration in the respective subscales.
Change from baseline in Affective Response to Exercise at 16 months | baseline and 16 months
  The Feeling Scale (FS) is an 11-point scale ranging from -5 ("Very bad") to +5 ("Very good"), which assesses the affective valence of exercise.
Change from baseline in Affective Response to Exercise at 4 months | baseline and 4 months
  The Feeling Scale (FS) is an 11-point scale ranging from -5 ("Very bad") to +5 ("Very good"), which assesses the affective valence of exercise.
Change from baseline in Affective Response to Exercise at 10 months | baseline and 10 months
  The Feeling Scale (FS) is an 11-point scale ranging from -5 ("Very bad") to +5 ("Very good"), which assesses the affective valence of exercise.
Change from baseline in Exercise Self-Efficacy at 16 months | baseline and 16 months
  The 9-item Modified Bandura's Exercise Self-Efficacy Scale will be used to measure how certain participants are/were that they would practice exercise under different conditions or restrictions. Scores range from 1 ("Very sure") to 4 ("Not at all sure"). Higher scores reflect lower exercise self-efficacy.
Change from baseline in Exercise Self-Efficacy at 4 months | baseline and 4 months
  The 9-item Modified Bandura's Exercise Self-Efficacy Scale will be used to measure how certain participants are/were that they would practice exercise under different conditions or restrictions. Scores range from 1 ("Very sure") to 4 ("Not at all sure"). Higher scores reflect lower exercise self-efficacy.
Change from baseline in Exercise Self-Efficacy at 10 months | baseline and 10 months
  The 9-item Modified Bandura's Exercise Self-Efficacy Scale will be used to measure how certain participants are/were that they would practice exercise under different conditions or restrictions. Scores range from 1 ("Very sure") to 4 ("Not at all sure"). Higher scores reflect lower exercise self-efficacy.
Self-regulation skills | 4 months (intervention's end), 10 and 16 months
  Action planning (i.e., when, where, what to do, and how often exercise) and coping planning (i.e., how to cope with setbacks and what to do to act according to one's intentions to exercise) will be assessed the Action Planning and the Coping Planning scales, comprising 5 items each. Action control will be measured with 6 items addressing its different facets, (i.e., self-monitoring, awareness of standards, and self-regulatory effort). Scores range from 1 ("Completely disagree") to 4 ("Totally agree"). Higher scores reflect greater self-regulation skills.
Perceived intervention climate | 4 months (intervention's end)
  Participants perception of the facilitators interpersonal behaviors will be measured with the Interpersonal Behaviors Questionnaire (IBQ), a 24-item instrument including three support subscales - perceived autonomy, competence, and relatedness support - and three thwarting subscales - perceived autonomy, competence, and relatedness thwarting. Scores range from 1 ("do not agree at all") to 7 ("completely agree"). Higher scores reflect greater support/thwarting in the respective subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Eliana V. Carraça, PhD, Principal Investigator — Universidade Lusófona, Faculdade de Educação Física e Desporto, Lisboa, Portugal
Locations (1):
- Universidade Lusófona, Campo Grande 376, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franco S, Carraca EV, Nobre I, Rodrigues B, Ilharco V, Kahlert L, Silva MN. Developing and testing the feasibility of a theory-based brief counseling intervention to promote physical activity in breast cancer survivors enrolled in the PAC-WOMAN trial. Pilot Feasibility Stud. 2025 Jan 11;11(1):4. doi: 10.1186/s40814-024-01587-0. PMID 39799368
- [Derived] Carraca EV, Rodrigues B, Franco S, Nobre I, Jeronimo F, Ilharco V, Gabriel F, Ribeiro L, Palmeira AL, Silva MN. Promoting physical activity through supervised vs motivational behavior change interventions in breast cancer survivors on aromatase inhibitors (PAC-WOMAN): protocol for a 3-arm pragmatic randomized controlled trial. BMC Cancer. 2023 Jul 5;23(1):632. doi: 10.1186/s12885-023-11137-1. PMID 37407950